CLINICAL TRIAL: NCT03923088
Title: Comparison Between Jacobson's Progressive Muscle Relaxation Technique and Audio-visual Distraction Technique in Reducing Dental Anxiety in Children During Dental Visit ; Randomized Clinical Trial
Brief Title: Comparison Between Jacobson's Progressive Muscle Relaxation Technique and Audio-visual Distraction Technique in Reducing Dental Anxiety in Children During Dental Visit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dina Hussien Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Dina Hussien Abdelhafez, principal investigator Dina Hussien Abdelhafez, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01234
Record Dates: First submitted 2019-04-16; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- jacobson's progressive muscle relaxation technique (Experimental)
  Interventions: Behavioral: jacobson's progressive muscle relaxation technique
- audiovisual distraction technique (Experimental)
  Interventions: Behavioral: audio-visual distraction technique
- conventional (No Intervention)

INTERVENTIONS:
Behavioral: jacobson's progressive muscle relaxation technique — This involves tensing specific muscle groups for 5-7 seconds, followed by 20 seconds of relaxation. The method can be demonstrated chairside, and should be practiced and rehearsed by the patient at home. Four major muscle groups are commonly tensed and relaxed. These are: 1) feet, calves, thighs, and buttocks; 2) hands, forearms, and biceps; 3) chest, stomach, and lower back; and 4) head, face, throat, and shoulders
  Arms: jacobson's progressive muscle relaxation technique
Behavioral: audio-visual distraction technique — audiovisual distraction not only leads to full involvement of scenes (visual and auditory), but it also induces a positive emotional reaction resulting in a relaxed experience.
  Arms: audiovisual distraction technique

SUMMARY:
Dental anxiety is fear associated with the thought of visiting the dentist for preventive care and dental procedures. Children with dental anxiety characterized by crying before dental checkup, tachycardia and aggressively clinging to the accompanying parent. It has been cited as the fifthmost common cause of anxiety by Agras et al. Dental anxiety may have major and long-lasting implications for the child and their family. Cohen et al reported that dental anxiety affects an individual's life in multiple ways. The physiological impacts included signs and symptoms of the fright response and feelings of exhaustion after a dental appointment, while the cognitive impacts included an array of negative thoughts, beliefs, and fears. Dental anxiety in children could remain a problem in adulthood if not handled properly thus it will affect oral health and psycho-social condition. This research is conducted to deliver different concepts in psychological and behavioral techniques in management of anxious pediatric dental patients.

ELIGIBILITY:
Inclusion Criteria:

* Children: 6 to 9 years old children. Teeth: tooth requiring dental treatment

Exclusion Criteria:

* Children having allergy to local anaesthesia or systemic problem. Refusal of participation Mentally ill or mentally retarded children

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
cooperation measured by modified venham rating scale | 1 hour
  Modified Venham rating scale provides details of positive and negative child's behavior. The scale ranges from total cooperation (0) to no cooperation (5)